CLINICAL TRIAL: NCT05828771
Title: Outcomes and Clinical Applications of Thin Free Flaps for Soft Tissue Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Mohamed Abdellatif, assistant lecturar at plastic surgery department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-Med-23-04-02MD
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: SOFT TISSUE DEFECTS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: THIN FREE FLAP — Flap design will be performed on the basis of the preoperative perforator mapping. Freestyle flap elevation will be performed under loupe magnification from one of the incisions until the perforators are reached

SUMMARY:
Flap coverage is often required to achieve primary wound closure and to achieve a good functional result. Free flap has gain popularity over random flap in soft tissue reconstruction to achive maximal cosmetic and functional outcome. Advances in reconstructive techniques have widened the application of free flap tissue transfer for repair of head and neck defects and have resulted in improved quality of life and both functional and aesthetic outcomes. Interference of high technology like CT Angio and Duplex ultra sound makes perforator detection more easy and more accurate. Fasciocutaneous free flaps raised in the traditional sub or supra-fascial planes can sometimes be thick and bulky. Elevating thin flaps has long been a goal of reconstructive surgeons. Thin flaps have numerous advantages in reconstruction. Thin flap is required in aesthetically significant areas, such as in fascial and hand reconstruction. In addition to their aesthetic importance, thin flaps are frequently required due to functional considerations. In head and neck reconstruction, bulky flaps may interfere with smooth swallowing and cause airway obstruction. In adition resurfacing of joint exposure require thin flap to maintain maximum joint function. Donor site shows better outcomes with thin free flap due to preservation of deep fatty layer that decrease the incidence of donor site neuroma and better countour when application of skin graft.

ELIGIBILITY:
Inclusion Criteria:

* All patients with soft tissue defects in different body regions who are prepared for free flap surgery. All patients under 65 year of age and above 5 years of age.

Exclusion Criteria:

* Patient who is not indicated for free flap. Patient above 65 year of age and below five year of age. Severely ill patient or with vascular problem or unfit for surgery.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
SUCEES RATE AND POTENTIAL COVERAGE | 6 months
  This study is designed for the clinical applications of thin free flaps regarding their coverage potential, dissection procedure and their outcomes (success and complications) as a reconstructive option

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Celik N, Wei FC, Lin CH, Cheng MH, Chen HC, Jeng SF, Kuo YR. Technique and strategy in anterolateral thigh perforator flap surgery, based on an analysis of 15 complete and partial failures in 439 cases. Plast Reconstr Surg. 2002 Jun;109(7):2211-6; discussion 2217-8. doi: 10.1097/00006534-200206000-00005. PMID 12045538
- [Background] Garg RK, Wieland AM, Hartig GK, Poore SO. Risk factors for unplanned readmission following head and neck microvascular reconstruction: Results from the National Surgical Quality Improvement Program, 2011-2014. Microsurgery. 2017 Sep;37(6):502-508. doi: 10.1002/micr.30116. Epub 2016 Sep 23. PMID 27658935
- [Background] Glass GE, Staruch RM, Sivakumar B, Stotland MA. Thin and superthin free flaps: An innovative approach to pediatric extremity reconstruction. J Plast Reconstr Aesthet Surg. 2022 Nov;75(11):3970-3978. doi: 10.1016/j.bjps.2022.06.090. Epub 2022 Jun 28. PMID 36163147
- [Background] Goh TLH, Park SW, Cho JY, Choi JW, Hong JP. The search for the ideal thin skin flap: superficial circumflex iliac artery perforator flap--a review of 210 cases. Plast Reconstr Surg. 2015 Feb;135(2):592-601. doi: 10.1097/PRS.0000000000000951. PMID 25357163